CLINICAL TRIAL: NCT00701870
Title: Phase 2 Randomized Study of Ezatiostat Hydrochloride (Telintra™, TLK199 Tablets) for Treatment of Chemotherapy Induced Neutropenia in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Receiving First-Line Chemotherapy
Brief Title: Study of Telintra for Treatment of Chemotherapy Induced Neutropenia in Patients With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study TLK199.2102 was terminated for lack of enrollment.
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TLK199.2102
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Chemotherapy induced neutropenia; CIN
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ezatiostat hydrochloride (Telintra®) (Experimental): Chemotherapy with docetaxel and carboplatin followed by Telintra until ANC recovery
  Interventions: Drug: ezatiostat hydrochloride (Telintra®)
- No Intervention (No Intervention): Chemotherapy with docetaxel and carboplatin alone

INTERVENTIONS:
Drug: ezatiostat hydrochloride (Telintra®) — 4500 mg orally per day in two divided doses
  Other Names: Telintra tablets; ezatiostat tablets
  Arms: ezatiostat hydrochloride (Telintra®)

SUMMARY:
TLK199.2102 was a multicenter Phase 2 randomized study to determine the effect of Telintra treatment on chemotherapy induced neutropenia (CIN) in patients with non small cell lung cancer receiving first-line therapy with carboplatin and docetaxel.

DETAILED DESCRIPTION:
TLK199.2102 was a multicenter Phase 2 randomized study to determine the effect of Telintra treatment on chemotherapy induced neutropenia (CIN) in patients with non small cell lung cancer receiving first-line therapy with carboplatin and docetaxel.

After randomization, patients in Treatment Arm 1, chemotherapy with carboplatin and docetaxel will be administered on Day 1 of each cycle, followed by Telintra at a starting dose of 3000 mg total daily dose (1500 mg orally, twice daily) on Day 2 until the absolute neutrophil count improves as confirmed by two consecutive measurement at least 24 hours apart. In Treatment Arm 2 (control arm), chemotherapy alone consisting of carboplatin and docetaxel will be administered on Day 1 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC
* Stage IIIb-Stage IV NSCLC
* ECOG performance status of 0-2
* Adequate liver and renal function
* Adequate bone marrow reserve

Exclusion Criteria:

* Treatment with neoadjuvant or adjuvant chemotherapy within 1 year
* Histologically confirmed mixed tumors containing small cell elements
* Treatment with radiotherapy (except limited in nature) within 3 weeks of randomization
* History of bone marrow transplantation or stem cell support
* Known history of CNS metastasis unless the patient has had treatment with surgery or radiotherapy, is neurologically stable and does not require oral or IV steroids or anticonvulsants
* History of HIV
* Grade 3 or 4 peripheral neuropathy
* Weightloss greater than 5% within 6 months
* Uncontrolled pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Duration of chemotherapy induced neutropenia | 6 weeks

SECONDARY OUTCOMES:
Duration of chemotherapy induced severe neutropenia | 6 weeks
Time to ANC recovery from ANC nadir | 6 weeks
Incidence of febrile neutropenia | 6 weeks
Incidence of G-CSF administration | 6 weeks
FACT-N quality of life assessment | 6 weeks
safety assessments | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail Brown, MD, Study Director — Telik
Locations (24):
- United States (24):
  - Central Hematology Oncology Medical Group, Alhambra, California
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Providence St. Joseph Medical Center, Burbank, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Wilshire Oncology Medical Group, La Verne, California
  - UCLA Medical Center, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Samsum Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Florida Hospital Cancer Institute, Ormand Beach, Florida
  - Suburban Hematology-Oncology Associates, PC, Lawrenceville, Georgia
  - Medical & Surgical Specialists, Galesburg, Illinois
  - Joliet Oncology/Hematology Associates, Ltd., Joliet, Illinois
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - Case Medical Center-University Hospitals, Cleveland, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Coastal Cancer Center, Myrtle Beach, South Carolina